CLINICAL TRIAL: NCT00113178
Title: Clinical Study to Evaluate the Safety and Efficacy of the CryoCor™ Cardiac Cryoablation System for the Treatment of Cavo-Tricuspid Valve Isthmus-Dependent Atrial Flutter
Brief Title: Safety and Efficacy of the CryoCor™ Cardiac Cryoablation System for the Treatment of Atrial Flutter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-AFL-02
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Flutter
Keywords: atrial flutter; cryoablation
MeSH Terms: conditions — Atrial Flutter

INTERVENTIONS:
Device: Catheter-based cardiac cryoablation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of right atrial intra-cardiac lesions created by transvenous catheter cryoablation in patients with atrial flutter.

DETAILED DESCRIPTION:
Catheter ablation of arrhythmias has become an accepted alternative to pharmacologic therapy. Cryoablation is a newer alternative to radiofrequency ablations. This study expands the prior pilot experience with the CryoCor™ Cardiac Cryoablation System to a larger cohort of patients with atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial flutter

Exclusion Criteria:

* Prior ablation
* Contraindication to intervention
* Poor general health

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Acute efficacy
Acute safety

SECONDARY OUTCOMES:
Long-term efficacy
Long-term safety

REFERENCES:
- See also: Related Info — http://www.cryocor.com/